CLINICAL TRIAL: NCT00864565
Title: Randomized, 2-way Crossover, Bioequivalence Study of Fentanyl 25 μg/h Transdermal System and Duragesic 25 μg/h Transdermal System Administrated as 1 x 25 μg/h Single Application in the Healthy Subjects
Brief Title: A Relative Bioavailability Study of Fentanyl 25 μg/h Transdermal System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 02348
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Fentanyl; Healthy subjects
MeSH Terms: interventions — Fentanyl; Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Fentanyl 25 μg/h transdermal system, single application
  Interventions: Drug: Fentanyl 25 μg/h transdermal system, single application
- B (Active Comparator): Duragesic 25 μg/h transdermal system single application
  Interventions: Drug: Duragesic 25 μg/h transdermal system single application

INTERVENTIONS:
Drug: Fentanyl 25 μg/h transdermal system, single application — A: Experimental Subjects received Corium International, Inc formulated products
  Other Names: Fentanyl
  Arms: A
Drug: Duragesic 25 μg/h transdermal system single application — B: Active comparator Subjects received Jassen Pharmaceutica Products, L.P. formulated products
  Other Names: Fentanyl
  Arms: B

SUMMARY:
To compare the rate and extent of absorption of fentanyl 25 μg/h transdermal system (test) and Duragesic (reference) administrated as 1 x 25 μg/h single transdermal system application.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, 2-period, 2-sequence, crossover design.

Official Title: Randomized, 2-way crossover, bioequivalence study of Fentanyl 25 μg/h transdermal system and Duragesic 25 μg/h transdermal system administrated as 1 x 25 μg/h single application in the healthy subjects

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be females and/or males, smokers and/or non-smokers, between 18 and 55 years of age.
* Subject capable of consent.
* Female subjects will be post-menopausal or surgically sterilized.

  1. Post-menopausal status is defined as absence of menses for the past 12 months or hysterectomy with bilateral oophorectomy at least 6 months ago.
  2. Sterile status is defined as hysterectomy, bilateral oophorectomy or tubal ligation at least 6 months ago.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C or HlV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 100 or over 140 mmHg, or diastolic blood pressure lower than 60 or over 90 mmHg; or heart rate less than 60 or over 100 bpm) at screening.
* Subjects with BMI >30.0.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than fourteen units of alcohol per week (1 Unit ≈ 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of abuse or dependency or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within I year of the screening visit.
* History of allergic reactions to fentanyl, naloxone or adhesives.
* History of allergic reactions to heparin.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO .inhibitors, neuroleptics, verapamil, quinidine) within 30 days prior to administration -of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* History or presence of any clinically significant liver or kidney disease or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug.
* Any history or presence of clinically significant neurological. endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Smoking more than 25 cigarettes per day.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical subinvestigator, contraindicates the subject's participation in this study.
* Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follows:

  1.less than 300 mL of whole blood within 30 days or 2.300 mL to 500 mL of whole blood within 45 days or 3.more than 500 mL of whole blood within 56 days .
* Subjects who have consumed food or beverages containing grapefruit (e.g. fresh, canned, or frozen) within 7 days prior to administration of the study medication.
* Subjects with a history or presence of asthma. chronic obstructive pulmonary disease or other pulmonary condition that may predispose to hypoventilation.
* Subjects with a history or presence of bradyarrythmias.

Additional criteria for females only:

* Breast-feeding subjects.
* Positive urine pregnancy test at screening (performed on all females).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2003-06; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 132 hours

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc, Québec, Quebec, Canada